CLINICAL TRIAL: NCT01635478
Title: A Prospective Observational Study of Assessment of Emergency Cancer Pain and Its Treatment Adequacy in Emergency Department of Tertiary Care Cancer Hospital.
Brief Title: A Observational Study of Assessment and Treatment Adequacy of Emergency Cancer Pain in Tertiary Cancer Hospital
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, DR. SWAPNIL YESHWANT PARAB, FELLOW, Tata Memorial Hospital
Other Study IDs: emcap2011
Record Dates: First submitted 2012-07-04; First posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: TO STUDY EMERGENCY CANCER PAIN PATTERNS AND TREATMENT ADEQUACY.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
EMERGENCY CANCER PAIN MANAGEMENT HAS BEEN INCONSISTENT AND INADEQUATE ACROSS THE GLOBE. THIS STUDY AIMS TO KNOW EMERGENCY ROOM CANCER PAIN PATTERNS AND TREATMENT ADEQUACY IN TERTIARY CARE CANCER HOSPITALS.

ELIGIBILITY:
Inclusion Criteria:

* ADULT CANCER PATIENTS REPORTING TO EMERGENCY ROOM WITH COMPLAINTS PRIMARILY OF PAIN

Exclusion Criteria:

* PATIENTS BELOW 18 YEARS OF AGE AND PATIENTS WITH INCOHERENT BEHAVIOUR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ADULT CANCER PATIENTS REPORTING TO EMERGENCY ROOM WITH COMPLAINTS PRIMARILY OF PAIN.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)